CLINICAL TRIAL: NCT00044317
Title: Health Effects of Particulate Acids in Late Adolescence
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8391-CP-001
Record Dates: First submitted 2002-08-26; First posted 2002-08-27 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: Airway Obstruction; Cough
Keywords: FEV; Smoking; antioxidents; lung growth
MeSH Terms: conditions — Airway Obstruction; Cough; Smoking

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This study was designed to follow a group of adolescents who were previously examined by questionnaire and pulmonary function tests when they were aged 8-10 years old. Approximately 50% of the population in 10 towns were seen again at age 17-18. Questionnaires and pulmonary function were repeated. The hypotheses being tested related to whether the previously seen levels of pulmonary function that were related to pollution levels in the towns persisted as the lungs of these children grew and whether dietary antioxidants influences level of attained pulmonary function.

ELIGIBILITY:
Children seen in a previous study at ages 8-10 from selected cities

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500